CLINICAL TRIAL: NCT04197596
Title: A Pilot Study in the Treatment of Refractory BK Infections With Related Donor BK Specific Cytotoxic T-cells (CTLs) in Children, Adolescents and Young Adult Recipients
Brief Title: Treatment of Refractory BK Infections With Related Donor BK Specific Cytotoxic T-cells (CTLs)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Nationwide Children's Hospital (Other); Johns Hopkins University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 590
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Viral Infection; Primary Immune Deficiency Disorder
MeSH Terms: conditions — Virus Diseases; Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BK CTL (Experimental): Eligible patients with refractory BK infection will receive up to 5 infusions of BK CTLs that are donor derived.
  Interventions: Biological: BK CTL

INTERVENTIONS:
Biological: BK CTL — Patient with refractory BK infection and a HLA Matched Related Donors: BK specific CTLs (2.5 x 104 CD3/kg) infused intravenously on day 0 and may be additionally reinfused at a minimum of every two weeks (depending on safety and efficacy) for a maximum of five total infusions (maximum 12.5 x 104 CD3/kg).
  Patients with refractory BK virus and a HLA Mismatched Related Donors: BK specific CTLs (0.5x104 CD3/kg) infused intravenously on day 0 and may additionally be reinfused at a minimum of every two weeks (depending on safety and efficacy) for a maximum of five total infusions (maximum 2.5 x 104 CD3/kg).

SUMMARY:
BK cytotoxic T cells (CTLs) manufactured with the Miltenyi CliniMACS Prodigy Cytokine Capture System will be safe and effective in decreasing specific viral load in children, adolescents and young adults (CAYA) with refractory BK infection post Allogeneic Hematopoietic Stem Cell Transplantation (AlloHSCT) or with primary immunodeficiencies (PID).

ELIGIBILITY:
Inclusion Criteria:

.1.1 Patients with refractory BK infection post allogeneic HSCT, post solid organ transplantation or with primary immunodeficiencies with either

* Increasing urine and/or plasma BK RT-PCR DNA (by 1 log) after 7 days or persistent quantitative qRT-PCR DNA copies after 14 days despite two weeks of appropriate anti-viral therapy AND/OR
* Medical intolerance to anti-viral therapies including:

  * 2 renal toxicity with cidofovir or other > grade 2 toxicities secondary to cidofovir And/or
* known resistance to cidofovir 1.2. Consent: Written informed consent given (by patient or legal representative) prior to any study-related procedures.

1.3 Performance Status > 30% (Lansky < 16 yrs and Karnofsky > 16 yrs) 1.4 Age: 0.1 to 79.99 years 1.5 Females of childbearing potential with a negative urine pregnancy test

Exclusion:

1. Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of BK CTL infusion
2. Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of BK CTL infusion
3. Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to BK CTL infusion
4. Thymoglobulin (ATG) or Alemtuzumab within 30 days
5. Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30%
6. Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory BK infection.
7. Any medical condition which could compromise participation in the study according to the investigator's assessment
8. Known HIV infection
9. Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.
10. Known hypersensitivity to iron dextran
11. Patients unwilling or unable to comply with the protocol or unable to give informed consent.
12. Known human anti-mouse antibodies

Ages: 1 Month to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 weeks
  Patients will be monitored for adverse events following each CTL infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided